CLINICAL TRIAL: NCT04622540
Title: A Prospective Randomized Controlled Trial for Application of External Biliary Drainage in Living Donor Liver Transplantation
Brief Title: EBD RCT Trial in Living Donor Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Suk Kyun Hong, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SNUHLT_EBD
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Liver Transplantation; Liver Transplant; Complications; Bile Stricture; Bile Leakage From Biliary Anastomosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Application of external biliary drainage
  Interventions: Procedure: External biliary drainage
- Control group (No Intervention): Conventional duct-to-duct anastomosis (with or without internal stent)

INTERVENTIONS:
Procedure: External biliary drainage — Application of external biliary drainage through duct-to-duct anastomosis
  Arms: Experimental group

SUMMARY:
This study was designed to demonstrate incidence of biliary complication rates after living donor liver transplantation according to the implantation of external biliary drainage throug duct-to-duct anastomosis site.

DETAILED DESCRIPTION:
Biliary complication is the most common complications after liver transplantation, and it happens more often after living donor liver transplantation (LDLT) than deceased donor liver transplantation.

Many transplant centers adopted their own methods to improve biliary complications after LDLT. One suggested method is the application of external biliary drainage (EBD).

A prospective study was planned to demonstrate effect of EBD on biliary complication after LDLT. Patients who underwent LDLT with duct-to-duct anastomosis will be randomly assinged to application of EBD or conventional duct-to-duct anastomosis without EBD according to a computer generated randomization sequence and allocated in a 1:1 ratio to one of two groups.

Primary outcome is biliary complication incidence 1 year after LDLT.

ELIGIBILITY:
Inclusion Criteria:

* Living donor liver transplantation
* Adult patient (>=18 years old)
* Patients who are available for at least 3 year follow-up after LDLT

Exclusion Criteria:

* Patients requring hepaticojejunostomy due to anatomical factor or underlying disease
* Re-transplantation
* Multiorgan transplantation
* Emergency transplantation

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of biliary complication within 1 year after LDLT | 1 year
  Biliary stricture/leakage

SECONDARY OUTCOMES:
Incidence of biliary complication within 3 year after LDLT | 3 year
  Biliary stricture/leakage
Complication associated with external biliary drainage | 3 year
  Dislocation, retraction, reposition, leakage through tube site, hemorrhage
Graft survival | 3 year
  Survival of liver graft
Patient survival | 3 year
  Patient survival after LDLT
Patient-reported outcome | 3 year
  Questionnaire survey

CONTACTS AND LOCATIONS:
Overall Officials: Suk Kyun Hong, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freise CE, Gillespie BW, Koffron AJ, Lok AS, Pruett TL, Emond JC, Fair JH, Fisher RA, Olthoff KM, Trotter JF, Ghobrial RM, Everhart JE; A2ALL Study Group. Recipient morbidity after living and deceased donor liver transplantation: findings from the A2ALL Retrospective Cohort Study. Am J Transplant. 2008 Dec;8(12):2569-79. doi: 10.1111/j.1600-6143.2008.02440.x. Epub 2008 Oct 24. PMID 18976306
- [Background] Akamatsu N, Sugawara Y, Hashimoto D. Biliary reconstruction, its complications and management of biliary complications after adult liver transplantation: a systematic review of the incidence, risk factors and outcome. Transpl Int. 2011 Apr;24(4):379-92. doi: 10.1111/j.1432-2277.2010.01202.x. Epub 2010 Dec 10. PMID 21143651
- [Background] Hwang S, Lee SG, Sung KB, Park KM, Kim KH, Ahn CS, Lee YJ, Lee SK, Hwang GS, Moon DB, Ha TY, Kim DS, Jung JP, Song GW. Long-term incidence, risk factors, and management of biliary complications after adult living donor liver transplantation. Liver Transpl. 2006 May;12(5):831-8. doi: 10.1002/lt.20693. PMID 16528711
- [Background] Jung DH, Ikegami T, Balci D, Bhangui P. Biliary reconstruction and complications in living donor liver transplantation. Int J Surg. 2020 Oct;82S:138-144. doi: 10.1016/j.ijsu.2020.04.069. Epub 2020 May 5. PMID 32387205
- [Background] Park CS, Jung BH, Hwang S, Park YH, Kang SH, Park GC, Song GW, Jung DH, Ahn CS, Kim KH, Moon DB, Ha TY, Lee SG. External biliary drainage in living donor liver transplantation using duct-to-duct anastomosis. Transplant Proc. 2014 Apr;46(3):678-81. doi: 10.1016/j.transproceed.2013.11.150. PMID 24767322
- [Background] Lee SG. A complete treatment of adult living donor liver transplantation: a review of surgical technique and current challenges to expand indication of patients. Am J Transplant. 2015 Jan;15(1):17-38. doi: 10.1111/ajt.12907. Epub 2014 Oct 30. PMID 25358749